CLINICAL TRIAL: NCT02505633
Title: A Randomized Comparison Between 1 Plane - 1 Injection (Cluster Approach) and 2 Plane - 2 Injection Ultrasound-guided Supraclavicular Brachial Plexus Block (US-SCBPB) in Upper Extremity Surgery
Brief Title: Comparison 1 Plane-1 Injection and 2 Plane-2 Injection Ultrasound-guided Supraclavicular Brachial Plexus Block
Acronym: US-SCBPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Mi Geum Lee, assistant professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: GBIRB2015-44
Record Dates: First submitted 2015-07-19; First posted 2015-07-22 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Radius Fractures
Keywords: brachial plexus block; nerve stimulator; ultrasound
MeSH Terms: conditions — Radius Fractures | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2P2I group (Experimental): subcutaneous injection is done widely. A nerve stimulating needle (Stimuplex insulated needle; D Plus B. Braun, Melsungen, Germany) attached to a nerve stimulator (Stimuplex HNS12; B. Braun, Melsungen, Germany) is advanced via an ultrasound in-plane approach. After the needle is penetrated the nerve sheath with a direction of downward, the nerve stimulator is then turned on. If hand muscle twitching is observed even at 0.3 mA, LA 15 mL (lidocaine mixed with epinephrine) is injected. After that, the stimulating needle is re-advanced at the behind site of the initial puncture site. And the needle is penetrated the nerve sheath with a direction of upward, and then the same process is performed and LA 15 mL is injected.
  Interventions: Device: Stimuplex insulated needle; Drug: lidocaine mixed with epinephrine
- 1P1I group (Active Comparator): After subcutaneous injection of 1 mL of 2% lidocaine, a nerve stimulating needle (Stimuplex insulated needle; D Plus B. Braun, Melsungen, Germany) attached to a nerve stimulator (Stimuplex HNS12; B. Braun, Melsungen, Germany) is advanced via an ultrasound in-plane approach from lateral to medial direction. After the needle is penetrated the nerve sheath, the nerve stimulator is then turned on, and the stimulation current starts at 0.5mA. If hand muscle twitching is observed even at 0.3 mA, local anesthetics 30 mL (lidocaine mixed with epinephrine) is injected.
  Interventions: Device: Stimuplex insulated needle; Drug: lidocaine mixed with epinephrine

INTERVENTIONS:
Device: Stimuplex insulated needle — 2P2I group: nerve stimulating needle is advanced twice and LA is injected 15 mL at a time.
  1P1I group: nerve stimulating needle is advanced once and LA is injected 30 mL.
  Other Names: (D Plus B.Braun)
Drug: lidocaine mixed with epinephrine — 2P2I group and 1P1I group use the same LA (1.5% lidocaine mixed with 1:200,000 epinephrine). But 2P2I group is injected LA at equally divided doses (15 mL at a time). 1P1I group is injected LA 30 mL at once.
  Other Names: 1.5% lidocaine mixed with 1:200,000 epinephrine

SUMMARY:
Ultrasound-guided supraclavicular brachial plexus block (US-SCBPB) has been a generalized regional anesthesia in upper extremity surgery. It is performed just above the clavicle, in which the neural cluster formed by the trunks or divisions of the brachial plexus is situated superolateral to the subclavian artery (SA).

In many approaches, corner pocket approach [deposit local anesthetic (LA) at the intersection of the SA, neural cluster, and the first rib] and cluster approach (direct deposit LA into the neural cluster after penetration of the sheath of brachial plexus) has been well known methods. And single or multiple injection techniques has been used with the above approaches.

DETAILED DESCRIPTION:
In clinical practices, the investigators observed that the neural cluster was shown differently every person on the ultrasound image. Some neural cluster is shown as a typical round cluster of grapes lateral to the SA, in which, any approaches of US-SCBPB can be possible and good success rates are anticipated. But in many cases, neural cluster was shown in part lateral or superolateral to the SA like slightly-hated SA on the ultrasound image, and it passes posterior to the SA when the probe follows the path of the neural cluster along the SA. In that case, corner pocket approach is hard to apply due to the position of the neural cluster far away from the first rib, cluster approach increases chance of lopsided spreading of the LA, and multiple injection is also hard to apply due to narrow-shaped neural cluster. Therefore, we hypothesized that double injection in different plane (we call this new approach as a 2 plane-2 injection approach) would achieve an effect of a "tridimensionally administered LA", which is presented like shortening the onset time or increasing rate of all four nerves block compared with the existing cluster approach (the investigators call this as an 1 plane- 1 injection approach in this study).

ELIGIBILITY:
Inclusion Criteria:

* all patients anticipating surgery of the wrist or hand with aged 18 to 80 years and an American Society of Anesthesiologists physical status (ASA) of I or II.

Exclusion Criteria:

* patients with preexisting neuropathy in the operated limb, ASA greater than III, coagulation disorders, known allergy to local anesthetics, local infection at the puncture site, chronic obstructive pulmonary disease or respiratory failure, pregnancy, breast-feeding and prior surgery in the supraclavicular region, BMI ≥ 35 kg/㎡, uncooperative patients and patients' refusal. an ultrasound view of the perfect circular neural cluster.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
rate of complete sensory blockade of all 4 nerves. | check 30 minutes after performing the block
  If the sensory on the site under the control of all 4 (median, radial, ulnar, musculocutaneous) nerves is checked as 0 (just feeling of touch or none ) separately, it is considered as a complete sensory block.
  the investigators compare the rate of complete sensory block with 2P2I group and 1P1I group.

SECONDARY OUTCOMES:
the onset time | check 30 minutes after performing the block
  The investigators compare the onset time (time required to obtain of a sensory block at the surgical incision site) with 2P2I group and 1P1I group.

CONTACTS AND LOCATIONS:
Overall Officials: Mi Geum Lee, MD, PhD, Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Department of Anesthesiology and Pain Medicine, Gachon University Gil Medical Center, Incheon, Guwol-dong, Namdong-gu, South Korea

REFERENCES:
- [Background] Techasuk W, Gonzalez AP, Bernucci F, Cupido T, Finlayson RJ, Tran DQ. A randomized comparison between double-injection and targeted intracluster-injection ultrasound-guided supraclavicular brachial plexus block. Anesth Analg. 2014 Jun;118(6):1363-9. doi: 10.1213/ANE.0000000000000224. PMID 24842181